CLINICAL TRIAL: NCT00524511
Title: A Comparative Study of Closure Techniques After Cesarean Section: Staples vs. Dermabond
Brief Title: Comparison Study of Wound Closure at Time of Cesarean Delivery: Dermabond Glue Versus Surgical Staples
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment, much data was missing as patients were lost to follow up
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Dawn Tasillo, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12462
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Cesarean Section
Keywords: cesarean; wound; Dermabond; superglue; staples; wound complications
MeSH Terms: conditions — Wounds and Injuries | interventions — Tissue Adhesives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Women receiving Dermabond for skin closure
  Interventions: Device: Surgical skin staples
- 2 (Active Comparator): Women receiving standard surgical skin staples
  Interventions: Device: Dermabond

INTERVENTIONS:
Device: Surgical skin staples — Standard method to close abdominal surgical wounds
  Arms: 1
Device: Dermabond — Alternative method (superglue) to close abdominal surgical wounds
  Other Names: Tissue adhesive
  Arms: 2

SUMMARY:
Women who have a cesarean delivery have a surgical incision on their abdomen (belly). The usual way to close this opening is with metal surgical staples. In many other types of surgery, surgical incisions are closed with a super-glue called Dermabond. The researchers at the University of Massachusetts believe Dermabond may be a safe alternative to using staples at the time of a cesarean delivery, but this has not been studied. Women who choose to participate will be randomly assigned to have the cesarean delivery skin incision closed with staples or Dermabond. The researchers will survey the patients to see how they felt about the experience and the appearance of their scar. The researchers will survey physicians performing the surgery to see how easy Dermabond was to use. The researchers will ask physicians to evaluate the appearance of the incision after a 6-week recovery period and will analyze complications (such as bruising, infection, or separation of the wound) in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing scheduled and non-scheduled cesarean deliveries

Exclusion Criteria:

* Prisoners
* Insulin-requiring diabetics
* Vertical skin incision
* Allergy to Dermabond

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn S Tasillo, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 4, 2007-July 9, 2010 Recruitment occured in the medical clinics and Labor and Delivery unit of an academic medical center
Pre-assignment Details: The study design dictates that patients be enrolled upon admission to Labor and Delivery. Subsequently, patients who did not deliver by cesarean delivery would be excluded
Groups:
- Group Receiving Alternative Skin Closure Method (Dermabond): Women receiving Dermabond for skin closure
- Group Receiving Standard Skin Closure Method (Surgical Staples: Women receiving standard surgical skin staples
Period: Overall Study
Arm/Group | Group Receiving Alternative Skin Closure Method (Dermabond) | Group Receiving Standard Skin Closure Method (Surgical Staples
Started | 68 | 68
Completed | 64 | 61
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Receiving Alternative Skin Closure Method (Dermabond) | Group Receiving Standard Skin Closure Method (Surgical Staples | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 67 | 68 | 135
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 68 | 136
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Wound Complication Rate
Description: Wound seroma or hematoma, wound separation, wound requiring packing, cellulitis, required extra medical clinic visits to evaluate wound
Time Frame: within six weeks of study intervention
Population: No participants were analyzed due to poor enrollment, subjects lost to follow-up and incomplete/partial data.
Arm/Group | Group Receiving Alternative Skin Closure Method (Dermabond) | Group Receiving Standard Skin Closure Method (Surgical Staples
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Satisfaction of Cosmesis of Surgical Wound
Description: survey questionnaire using a visual analog scale to inquire about incision appearance, satisfaction with method of closure and comparison to previous closure type (if applicable)
Time Frame: before hospital discharge after surgery
Population: No participants were analyzed due to poor enrollment, subjects lost to follow-up and incomplete/partial data.
Arm/Group | Group Receiving Alternative Skin Closure Method (Dermabond) | Group Receiving Standard Skin Closure Method (Surgical Staples
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group Receiving Alternative Skin Closure Method (Dermabond) | Group Receiving Standard Skin Closure Method (Surgical Staples
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes